CLINICAL TRIAL: NCT03650855
Title: Vertebral Bone Quality and Prediction of Screw Loosening in Spine Fusion
Acronym: QOAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17046J
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-03

CONDITIONS: Spine Fusion for Degenerative Spine Disease
Keywords: degenerative spine disease; screw loosening; Quantitative CT scan; vertebral bone density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Finding a way to use Vertebral CT scan will help to predict screw loosing risk in spinal fusion for degenerative spine disease. Patients who will undergo at least two spine fusion levels for degenerative spine disease will be enrolled in. Before surgery, patients will undergo a spinal QCT scan with a calibrated phantom. The calibrated bone density, at bone-implant interface, will be assessed using dual energy CT scan immediately after surgery, and six months later. The primary outcomes will be the difference between the two values of the bone implant interface. The difference between density values will be correlated to the pre-op bone density value.

DETAILED DESCRIPTION:
Screw loosening is a real problem in degenerative spine surgery because of the morbidity of secondary surgery sometimes needed for elderly patients. Today, there is no real possibility to know before surgery if cemented screws are needed or not. The use of cemented screws has its morbidity. In fact, bone densitometry is not a good exam to predict the bone quality in degenerative spine because of the arthritis. T-score in degenerative spine can be overestimated. The goal of our study is analyze the bone-implant interface after spine fusion using dual-energy CT scan technology which can provide pictures without artifact compared to standard CT scan. This is a prospective observational monocentric study. Patients over 18 years old and have undergone at least two primary spine fusion levels will be enrolled. The exclusion criteria are the use of cemented screws, secondary surgery and neurodegenerative disease. The primary outcome will be the change in the bone-implant interface at six months post-surgery compared to the interface after surgery. The change will be assessed by calibrated dual CT scan. The interface bone density will be assessed using calibrated scans, and correlate to the true vertebral bone density measured before surgery with a QCT. We hope that this study can provide a simple and reproducible help for surgeons to choose between uncommented and cemented screws for their spine fusions surgeries.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* needed a minimum 2 levels spinal fusion
* agreed protocol

Exclusion Criteria:

* Cimented pedicular screws
* secondary surgery
* neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by their surgeon during the current consultation 3 months before the surgery where the decision must support an arthrodesis of at least 2 levels between T3 and S1. The surgeon checks the inclusion criteria and offers the patient to participate. Inclusion will be done during this consultation. Patients will be informed by the surgeon of the nature of the study. They are intended to provide information to this effect and a certificate of non-opposition to the participation will be.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Change of bone-implant interface at 6-month follow up compared to post operative interface assessed on Dual energy CT Scan | 6 montths
  Assessment of bone-implant interface (1 to 3 mm around the screw) using calibrated bone density on spinal dual energy CT scan just after surgery and at 6 months of follow up. Comparison between the two measured values.

SECONDARY OUTCOMES:
evolution of bone density of non instrumented levels between T0 and 6 months follow up assessed with Dual Energy CT scan | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugues HM PASCAL-MOUSSELARD, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No